CLINICAL TRIAL: NCT03171948
Title: Effects of a Limited Almond Consumption After a Successful Weight Loss by a Comprehensive Weight Loss Plan on Weight Maintenance in Healthy Obese Female Adults: a Randomised Clinical Trial
Brief Title: Effects of a Limited Almond Consumption After a Weight Loss Plan on Weight Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-205
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Overweight
Keywords: almond; weight loss; Weight maintenance; hypoenergetic diet
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — SEMA7A protein, human

STUDY DESIGN:
Intervention Model Description: Almond Group (AG) are asked to have a 30 gr. almond every day in their afternoon snack plus following the hypoenergetic diet Nut Free group (NFG), as control group, who continue their diet without any nut consumption.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond group (Experimental): Almond Group (AG) are asked to have a 30 gr. almond every day in their afternoon snack plus following the hypoenergetic diet
  Interventions: Behavioral: Almond Group
- Nut Free group (Experimental): Nut Free group (NFG), as control group, who continue their diet without any nut consumption.
  Interventions: Behavioral: Nut Free group

INTERVENTIONS:
Behavioral: Almond Group — Almond Group (AG) are asked to have a 30 gr. almond every day in their afternoon snack plus following the hypoenergetic diet
  Other Names: AG group
  Arms: Almond group
Behavioral: Nut Free group — continue their diet without any nut consumption.
  Other Names: NFG
  Arms: Nut Free group

SUMMARY:
The purpose of this study is to assess the effects of limited portion of almond consumption after a successful weight loss by a comprehensive weight loss plan (NovinDiet Plan) on weight maintenance in obese female adults.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18-45 years of age.
* Body mass index (BMI) between 23-30 kg/ m² who lost at least 10% of her initial weight by the diet plan.
* Must be able to have moderate exercise.
* Must be interested to keep weight loss.

Exclusion Criteria:

* No Allergy to nut products
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next 6 months.
* Taking medications that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
weight loss | 6 Month
  kg

SECONDARY OUTCOMES:
Waist circumference | 6 Month
  cm
Fasting blood glucose | 6 Month
  mmol/l
Fasting insulin level | 6 Month
  mU/l
HbA1c | 6 Month
HOMA-IR | 6 Month
  percentage (%)
lipid profiles | 6 Month
  mmol/l
liver function | 6 Month
  U/l

CONTACTS AND LOCATIONS:
Locations (1):
- NovinDiet Clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided